CLINICAL TRIAL: NCT01989611
Title: Implementation of the Pre-Exposure Prophylaxis (PrEP) to HIV: A Demonstrative Project.
Acronym: PrEPBrasil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: University of Sao Paulo (Other); Centro de Referência e Treinamento DST/Aids (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PrEP Brasil; 08405912.9.1001.5262 (Registry Identifier: CAAE - Plataforma Brasil - IPEC / FIOCRUZ)
Record Dates: First submitted 2013-10-30; First posted 2013-11-21 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: HIV
MeSH Terms: interventions — Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- emtricitabine / tenofovir 200/300 mg (Other): Fixed dose combination of emtricitabine / tenofovir 200/300 mg once daily orally during one year.
  Interventions: Drug: emtricitabine / tenofovir 200/300 mg

INTERVENTIONS:
Drug: emtricitabine / tenofovir 200/300 mg — Fixed dose combination of emtricitabine / tenofovir 200/300 mg once daily orally during one year
  Other Names: Truvada

SUMMARY:
A prospective, open, multicenter,demonstrative of PrEP, which aims to assess the acceptability, feasibility and safety from chemoprophylaxis co-formulated emtricitabine / tenofovir disoproxil fumarate (FTC / TDF) administered orally, once daily, to MSM and transgender women . The demonstration project aims to include 400 participants over 12 months, with 200 at IPEC-Fiocruz, 100 at CRT-SP and 100 at USP.

DETAILED DESCRIPTION:
Subjects preliminarily eligible who choose to receive PrEP will be included after obtaining the informed consent and confirmation of eligibility within 45 days after the screening visit.

Once included, participants will be examined in a follow-up visit performed four weeks later and evaluated for evidence of seroconversion to HIV, medication compliance and clinical toxicity. The second follow-up visit will occur at 12th week and every 12 weeks successively (quarterly). Quarterly visits include HIV testing, serum creatinine and counseling on medication compliance and risk reduction.

The study has a total of 6 visits. In all visits will be assessed the risks, HIV testing will be performed, monitoring of renal function and dispensing of the drug Truvada [emtricitabine 1 tablet (FTC) / tenofovir (TDF) (200/300 mg) once a day orally for 12 months].

Participants who have completed 12 months of follow-up or prematurely discontinue a PrEP will be encouraged to return for a follow-up visit after discontinuation of medication for monitoring of the status and evaluation of HIV as the resolution of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Male (at birth);
* Willing and able to provide informed consent in writing;
* Age = or > 18 years;
* not infected by HIV-1, in accordance with the flowchart of testing from Brazilian Ministry of Health;
* Evidence risk for acquiring HIV-1, including any of the following:

  1. Anal sex without a condom with two or more men or transgender women in the last 12 months, or
  2. 2 or more episodes of anal sex with at least one partner HIV + in the last 12 months, or
  3. Sex with a man or trans woman and diagnosis of any of the following STDs in the last 12 months: syphilis, rectal gonorrhea or chlamydial infection in the rectum.
* Able to provide a residential address or contact phone itself, or two personal contacts who would know about his whereabouts during the study period demonstrative;
* Adequate renal function: Creatinine clearance > or = 60 ml / min, estimated by the formula modification of diet in renal disease (MDRD, from English 'Modification of Diet in Renal Disease') within 45 days of enrollment;
* urine Tape with negative result or showing only traces of protein within 45 days prior to enrollment;

Exclusion Criteria:

* Signs or symptoms of acute HIV infection,which is confirmed by laboratory examination in subsequent samples;
* Active and severe infections previously diagnosed, including active tuberculosis or osteomyelitis and all infections requiring parenteral antibiotics (except STD that require intramuscular injections of antibiotics);
* clinically significant active medical problems, including heart disease poorly controlled (eg, symptoms ischemia, congestive heart failure) previously diagnosed malignancy, or which will require additional treatment;
* Patients with positive tests for antigens of hepatitis B surface (HBsAg);
* History of pathological bone fractures unrelated to trauma;
* Patients using any of the following: ARV, including nucleoside inhibitors, non-nucleoside reverse transcriptase inhibitors, protease inhibitors and antiretroviral agents under study, treatment with interferon (alpha, beta, or gamma) or interleukin (e.g. ,IL-2), with potential significant nephrotoxic agents, other agents which may inhibit or compete for renal elimination via active tubular secretion (eg probenecid) and / or other agents under study;
* Participation in a clinical trial using concomitant agents under investigation, including placebo-controlled trials using such agents;
* Patients who have any condition at the time of inclusion in the study, according to the opinion of the investigator, may prevent the provision of informed consent, make study participation unsafe, complicate data interpretation, or interfere anyway with the achievement of project objectives.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Different compliance evaluations (the measure is a composite - please see description) | two years
  Acceptance and refusal rates Correlation of socio-demographic factors of acceptance and refusal Duration of PrEP Side effects and toxicities, including elevations of creatinine Adherence to PrEP: number of tablets per day, patterns of adherence Number of male sexual partners, by serostatus and condom use, and episodes of anal sex by partner serostatus, the interviewee practices and condom use.

SECONDARY OUTCOMES:
Number of patients infected and relation with medication compliance (the measure is a composite - please see description) | two years
  Knowledge about PrEP Reasons for the choice and refusal of PrEP seroconversions rate Patterns of resistance to anti-HIV among people who become infected Self-reports of deviation (selling or sharing) of PrEP medication Space needs and staff social harm Prevalence of sexually transmitted diseases

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Grinsztejn, PhD, Principal Investigator — Instituto de Pesquisa Clínica Evandro Chagas - Fiocruz
Locations (3):
- Brazil (3):
  - Instituto de Pesquisa Clínica Evandro Chagas - IPEC / FIOCRUZ, Rio de Janeiro, Rio de Janeiro
  - Centro de Referência e Treinamento DST/AIDS, São Paulo, São Paulo
  - University of Sao Paulo - Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo

REFERENCES:
- [Derived] Marins LMS, Torres TS, Leite IDC, Moreira RI, Luz PM, Hoagland B, Kallas EG, Madruga JV, Liu AY, Anderson PL, Grinsztejn B, Veloso VG. Performance of HIV pre-exposure prophylaxis indirect adherence measures among men who have sex with men and transgender women: Results from the PrEP Brasil Study. PLoS One. 2019 Aug 20;14(8):e0221281. doi: 10.1371/journal.pone.0221281. eCollection 2019. PMID 31430318
- [Derived] Grinsztejn B, Hoagland B, Moreira RI, Kallas EG, Madruga JV, Goulart S, Leite IC, Freitas L, Martins LMS, Torres TS, Vasconcelos R, De Boni RB, Anderson PL, Liu A, Luz PM, Veloso VG; PrEP Brasil Study Team. Retention, engagement, and adherence to pre-exposure prophylaxis for men who have sex with men and transgender women in PrEP Brasil: 48 week results of a demonstration study. Lancet HIV. 2018 Mar;5(3):e136-e145. doi: 10.1016/S2352-3018(18)30008-0. Epub 2018 Feb 18. PMID 29467098